CLINICAL TRIAL: NCT04474366
Title: The Effect of Pectoral Blocks on Perioperative Pain in Simple Mastectomy and Breast Reduction in Gender Affirmation Surgery
Brief Title: The Effect of Pectoral Blocks on Perioperative Pain in Gender Affirmation Top Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-28267
Record Dates: First submitted 2020-06-29; First posted 2020-07-16 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Gender Dysphoria; Opioid Use; Pain, Postoperative
MeSH Terms: conditions — Gender Dysphoria; Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline (Sham Comparator): Control group will receive an injection of 20ml of saline between the pectoralis minor and serratus anterior muscles bilaterally and 10ml of saline between the pectoralis minor and pectoralis major muscles bilaterally.
  Interventions: Other: Saline (0.9%)
- Ropivacaine (Experimental): Intervention group will receive an injection of 20ml of 0.2% Ropivacaine between the pectoralis minor and serratus anterior muscles bilaterally and 10ml of 0.2% Ropivacaine between the pectoralis minor and pectoralis major muscles bilaterally (Not to exceed 225mg or 3.5mg/kg).
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — Ropivacaine 0.2% Injectable Solution injected as part of the Pectoralis Nerve Block
  Arms: Ropivacaine
Other: Saline (0.9%) — Saline injection as sham block in identical fashion as Pectoralis Nerve Block
  Arms: Saline

SUMMARY:
Despite recent advancements with regional and local anesthesia, postoperative pain continues to be a major concern for patients undergoing breast surgery. Opioids, often in combination with NSAIDS and/or gabapentioids, have been the main pharmacologic pain control strategy in the postoperative period. The pectoral nerve block is a regional anesthetic technique, which is effective at providing postoperative anesthesia in breast surgeries. However, this has only been studied in oncologic-related breast operations. It is our aim to study the effects of pectoral regional nerve blocks in patients undergoing breast reduction for gender affirmation. The overall goal is to establish an effective pain control regimen utilizing regional anesthetic techniques in this patient population. The specific objective of this proposal is to evaluate the effectiveness of these blocks on perioperative and postoperative analgesia. The hypothesis is that participants undergoing gender-affirmation breast surgery who receive a pectoral nerve block will have less perioperative and postoperative pain as well as reduced opioid consumption compared to those receiving a placebo. Participants who are undergoing gender affirmation breast reduction surgery will be randomized to either receive a preoperative nerve block or to receive a placebo. Intraoperative and postoperative opioid requirements will be compared in addition to post-operative pain scores. Participants will be asked to fill out a pain diary during their first week postoperatively. They will also be asked to document if, and when, narcotic pain medication was required for pain control. The two groups will be compared to determine if there was any difference in pain scores as well as narcotic medication requirements.

DETAILED DESCRIPTION:
All participants will be seen in clinic with the attending surgeon anywhere from two weeks to a few months prior to the date of surgery. Participants will also have a pre-op visit with anesthesia a few weeks before surgery. They will undergo a standard anesthesia preoperative evaluation, which will include a medical chart review, physical exam, and appropriate laboratory studies. The preoperative evaluation will be identical for those participating in the study and those who do not. If no contraindications to the Pectoralis Nerve Block (PECS I and II block) are identified by the surgeon and/or anesthesiologist, participants will be approved to participate. The participants will be introduced to the study either during their clinic visit prior to surgery or over the telephone a few days prior to surgery. All questions will be answered by one of the study investigators. A study consent will be obtained from the participants and they will then will be randomized into either control (sham block) or experimental (PECS I and II block) group.

On the day of surgery, as per standard of care, each participant will undergo a general anesthetic in the same manner with conventional perioperative management. During induction of anesthesia, up to 2mg of midazolam and/or up to 100mcg of fentanyl will be given. The above protocol will be followed regardless of study participation and study group (if participating). After induction of anesthesia, the nerve blocks, or control blocks, will be performed. The regional anesthesia team will be involved in all patients, whether in the control or intervention group. All patients will be come and go regardless of group.

Group 1 (control) will receive an injection of 20ml of saline between the pectoralis minor and serratus anterior muscles bilaterally and 10ml of saline between the pectoralis minor and pectoralis major muscles bilaterally.

Group 2 (treatment) will receive an injection of 20ml of 0.2% Ropivacaine between the pectoralis minor and serratus anterior muscles bilaterally and 10ml of 0.2% Ropivacaine between the pectoralis minor and pectoralis major muscles bilaterally. (Not to exceed 225mg or 3.5mg/kg).

PECS I and II Block Technique: Performed in the supine position with the arms abducted 90 degrees at the shoulder. Using an ultrasound transducer in the parasagittal plane, the axillary artery and vein are identified just inferior to clavicle and medial to coracoid process. Additionally, the 2nd rib is identified and the transducer is slid inferiorly until the 3rd and 4th rib are identified. At this point the pectoralis major, minor, and serratus anterior muscles are seen. Then the block needle is inserted through the skin and advanced into the fascial plane between pectoralis minor and serratus anterior muscles. After negative aspiration, the anesthetic is injected into the plane watching for hydrodissection of the muscles. A total volume of 20ml is injected. Then the needed is withdrawn until the tip is located in the fascial plane between the pectoralis major and minor muscles. 10ml of anesthetic is injected into this plane.

General anesthesia is maintained in the standard fashion. The anesthesiologist will administer Fentanyl as he or she feels necessary during the operation. Post operatively, in the PACU, participants will be given IV hydromorphone as needed for pain. Pain scales will be documented at set time points post operatively and participants will be given pain diaries to document these pain scores as well as their opioid consumption. All patients will be sent home with a prescription for 20 tablets of Norco 5mg/325mg. Participants will be asked to document their pain scores at the following post op time points: 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 48 hours, 72 hours, 1 week. Participants will return their pain diaries at the 1 week post operative visit. This visit is a standard of care follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I-III
* Ages 18-65
* Undergoing gender confirmation breast reduction surgery by a single surgeon at a single center

Exclusion Criteria:

* Previous breast surgeries
* Current breast cancer or history of treatment for breast cancer
* Current chronic pain syndromes
* Coagulopathy
* Allergy to local anesthetics
* Infection at the injection site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Kim, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. For any purpose.

REFERENCES:
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] M N, Pandey RK, Sharma A, Darlong V, Punj J, Sinha R, Singh PM, Hamshi N, Garg R, Chandralekha C, Srivastava A. Pectoral nerve blocks to improve analgesia after breast cancer surgery: A prospective, randomized and controlled trial. J Clin Anesth. 2018 Mar;45:12-17. doi: 10.1016/j.jclinane.2017.11.027. Epub 2017 Dec 11. PMID 29241077
- [Background] Benotsch EG, Zimmerman R, Cathers L, McNulty S, Pierce J, Heck T, Perrin PB, Snipes D. Non-medical use of prescription drugs, polysubstance use, and mental health in transgender adults. Drug Alcohol Depend. 2013 Sep 1;132(1-2):391-4. doi: 10.1016/j.drugalcdep.2013.02.027. Epub 2013 Mar 17. PMID 23510637
- [Background] Day JK, Fish JN, Perez-Brumer A, Hatzenbuehler ML, Russell ST. Transgender Youth Substance Use Disparities: Results From a Population-Based Sample. J Adolesc Health. 2017 Dec;61(6):729-735. doi: 10.1016/j.jadohealth.2017.06.024. Epub 2017 Sep 21. PMID 28942238
- [Derived] Wallace AB, Song S, Yeh P, Kim EA. The Effect of Pectoral Nerve Blocks on Opioid Use and Postoperative Pain in Masculinizing Mastectomy: A Randomized Controlled Trial. Plast Reconstr Surg. 2024 Mar 1;153(3):570-577. doi: 10.1097/PRS.0000000000010707. Epub 2023 May 23. PMID 37220393

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline | Ropivacaine
Started | 23 | 27
Completed | 21 | 22
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Ropivacaine | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (8.7) | 27.1 (7.2) | 27.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 22 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Post Operative Pain Scores
Description: Participant recorded Numerical Rating Scale (NRS) pain scores post operatively. Scale ranges from 0 to 10. 0 represents no pain at all. 10 represents most severe pain.
Time Frame: 1 week post operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline | Ropivacaine
Number analyzed (Participants) | 22 | 21
score on a scale | 3.0 (1.8) | 3.6 (1.6)

2. Secondary Outcome: Comparison of Intra Operative Narcotic Requirements
Description: Intraoperative narcotic administration will be compared. Narcotic administration will be acquired through chart review. Total dose of IV hydromorphone intraoperatively will be collected.
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents
Arm/Group | Saline | Ropivacaine
Number analyzed (Participants) | 21 | 22
Morphine Milligram Equivalents | 11.1 (3.5) | 9.8 (4.5)

3. Secondary Outcome: Comparison of Post Operative Narcotic Requirements
Description: Self reported narcotic intake postoperatively. Number of pills taken will be recorded. Each group's number of pills will be averaged.
Time Frame: 1 week post operative
Measure: Median (Inter-Quartile Range); unit: Morphine Milligram Equivalents
Arm/Group | Saline | Ropivacaine
Number analyzed (Participants) | 21 | 22
Morphine Milligram Equivalents | 40.0 [15 to 65] | 37.5 [15.4 to 71.7]
Statistical Analysis 1: Comparison: Saline vs Ropivacaine; Test type: Superiority; p = 0.72, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Subjects were followed post operatively at designated time points after the surgery. These included 1 week, 2 weeks, 6 weeks, 3 months, and 6 months. Any adverse event encountered in this time frame was reported
Arm/Group | Saline | Ropivacaine
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04474366/Prot_SAP_000.pdf